CLINICAL TRIAL: NCT07056894
Title: Evaluating a Brief Virtual Cognitive Remediation Therapy Intervention for Those With Early Phase Psychosis and Substance Misuse in NS/NL: Addressing Challenges in Underserviced Areas
Brief Title: Effects of Action-Based Cognitive Remediation on Substance Misuse in Early Phase Psychosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Canadian Research Initiative in Substance Misuse (Other)
Responsible Party: Principal Investigator, Phil Tibbo, Principal Investigator, Nova Scotia Health Authority
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 74209
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Psychosis; Alcohol Use Disorder; Cannabis Use Disorder
Keywords: alcohol; cannabis; action based cognitive remediation; psychosis
MeSH Terms: conditions — Psychotic Disorders; Alcoholism; Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: 50 participants will choose either treatment as usual in an Early Intervention for Psychosis Service (EIS with 1 hour of psychoeducation or EIS plus Action-Based Cognitive Remediation for alcohol/cannabis misuse.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (No Intervention): Standard early intervention care and one psychoeducation session on the impacts substance use on recovery from psychosis.
- Action-Based Cognitive Remediation (ABCR) (Experimental): Action-Based Cognitive Remediation with an aim to reduce alcohol and/or cannabis consumption
  Interventions: Behavioral: Action-Based Cognitive Remediation

INTERVENTIONS:
Behavioral: Action-Based Cognitive Remediation — ABCR is a 16 session intervention involving computer-based drills, real-life simulations, and therapist-facilitated discussions intended to promote cognitive strategy monitoring and transfer of cognitive strategies to daily life. The sessions cover the follow key topics: Speed & Attention, Memory, Executive Functioning, and Social Cognition.
  Arms: Action-Based Cognitive Remediation (ABCR)

SUMMARY:
Psychotic disorders impact 4.6 people per 1000 globally, with approximately 1.5 million Canadians affected. The age of onset for psychotic disorders often begin during the critical years of youth and early adulthood, resulting in significant challenges for individuals and their families, including difficulties with thinking, relationships, and overall well-being. They also carry significant economic costs, both for health care and lost productivity. Early intervention services have been shown to improve outcomes when provided during the first few years of illness known as early phase psychosis (EPP). However, substance use, especially alcohol and cannabis, can interfere with the effectiveness of these services. Many young people with psychosis misuse these substances, which can harm brain development, worsen symptoms, reduce medication use, and lower quality of life. Despite understanding the risks, there are few effective ways to reduce substance misuse in patients with EPP.

One promising approach to reducing substance misuse in this population is cognitive remediation therapy, which helps improve thinking skills and everyday functioning. Studies have found that some cognitive remediation therapies can help reduce alcohol use in chronic schizophrenia, but there is limited research targeting the EPP population. Our research team at the Nova Scotia Early Psychosis Program recently completed a pilot study that indicated a therapy called Cognitive Enhancement Therapy (CET) helped participants reduce their problematic alcohol and cannabis use. However, challenges with recruitment and lower attendance rates noted towards the end of the 6-month therapy course suggests that patients with EPP would benefit more from a therapy with a shorter timeframe. Alternatively, Action-Based Cognitive Remediation (ABCR) targets the same cognitive domains believed to help reduce substance use as CET, but has a shorter, more concise schedule. ABCR cover 16 sessions delivered bi-weekly for 2 months, compared to 45 sessions over 6 months of CET. ABCR has been tested in the EPP population and has shown positive results when delivered in person, hybrid and remotely. Although this therapy is demonstrating benefits for patients including improvement in daily functioning and social cognition, its effects on substance misuse have not been researched. This study aims to investigate whether treatment with ABCR helps patients with EPP reduce their alcohol and/or cannabis use.

DETAILED DESCRIPTION:
Subjects will be recruited from the provincial Early Psychosis Intervention Nova Scotia programs (with the central site located in Halifax at the Nova Scotia Early Psychosis Program) and the Psychosis Intervention Early Recovery program in St. John's, Newfoundland. This is an open choice clinical trial comparing Action-Based Cognitive Remediation (ABCR) to treatment as usual (TAU) in early phase psychosis subjects. Following screening procedures, the participants will be offered the choice to enroll in the intervention or TAU group. Those who select ABCR will attend 16 bi-weekly therapy sessions over 2 months in a virtual group format. The TAU group will involve involved one brief psychoeducation session on the impacts of substance use in general on recovery.

This study will collect four different types of variables: demographic (things that describe the participants), clinical (things that describe how ill the individuals are), substance use (things that measure how much or how reliant participants are on recreational substances), and neuropsychological (things that measure cognitive functioning such as attention, memory, verbal learning, and executive functioning). These variables will be collected at baseline, 2 months (therapy end), and 3 months post-therapy for both the intervention and TAU group.

Demographic variables: Age, sex, gender, ethnicity, highest education level attained and current employment or education status as well as religious status (observing/not observing/do not identify) will be collected at baseline. Employment and school enrollment will be measured again at the end of the intervention. Relationship and living status will also be collected at baseline and end of the intervention.

Current medications will be recorded as there is some debate on the possible impact of some antipsychotic and antidepressant medications on reducing alcohol and cannabis use. Health resource utilization will include hospitalizations, number of missed clinical appointments with the EIS and emergency room visits for the trial period. All of which can be obtained from the patient's clinician.

Substance use variables: A contemplation ladder tool focused on alcohol and/or cannabis use will be used at baseline to assess willingness to change substance use to explore if readiness to change influences engagement with treatment and outcomes. The remaining measurements will be used at the three specified time-points. The Cannabis Use Disorder Identification Test - Revised (CUDIT-R) will collect data on hazardous cannabis use. The WHO Alcohol, Smoking and Substance Involvement Screening Test (WHO-ASSIST) will be administered to screen for all substance use including tobacco, alcohol and other recreational and illicit substances. The Timeline Follow-back (TLFB) method will collect detailed information about the last 30 day use of alcohol and/or cannabis. The alcohol use TLFB will collect the number of drinks consumed on each day. The cannabis use TLFB will collect information on cannabis quantity (gm/day), frequency (e.g. daily, times/week), type of product used (e.g. dried flower, concentrates, edibles) and potency (e.g. THC %, THC/CBD). Potency data will be self-report though also explored through websites used for product purchase.

Clinical variables: The Positive and Negative Symptom Scale (PANSS) will measure negative and positive psychotic symptom severity. Overall psychosis symptoms will be measured by the Clinical Global Impression scale, for both severity and improvement (CGI-S, CGI-I). The World Health Organization Disability Assessment Schedule 2 (WHODAS 2.0) will measure functioning across cognitive, mobility, self-care, getting along, life activities, and participation domains. The Calgary Depression Scale for Schizophrenia (CDSS) will assess the level of depression, and the Beck Anxiety Inventory (BAI) will examine anxiety symptoms.

Neuropsychological profile: The Digit Vigilance Test (DVT) will measure attention during a rapid visual tracking task. The California Verbal Learning Test 3 (CVLT3) will measure episodic verbal learning including verbal learning, immediate memory, and delayed memory. Trail Making Test A (TMT-A) will measure processing speed and the Trail Making Test B (TMT-B) will identify deficits in executive functioning. The Mayer-Salovey-Caruso Emotional Intelligence Test (MSCEIT) will provide a social cognition composite score.

ELIGIBILITY:
Inclusion Criteria:

* This study will enroll individuals 16-30 years of age from the Early Intervention Services for Psychosis programs in Nova Scotia and the Psychosis Intervention Early Recovery program in Newfoundland
* Diagnosed with a primary psychotic disorder (e.g. schizophrenia, schizoaffective disorder, and unspecified schizophrenia spectrum disorder)
* Less than 5 years of psychotic illness
* Has problematic alcohol and/or cannabis use (score of 8 or higher on the World Health Organization Alcohol Use Disorders Identification Test (WHO-AUDIT) or Cannabis Use Disorder Identification Test-Revised (CUDIT-R)).

Exclusion Criteria:

* Current stimulant use disorder

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in cannabis consumption | Baseline, 2 months, 5 months
  Cannabis Timeline Followback (TLFB) is a retrospective past 30 day calendar method used to collect detailed information about current cannabis use, which includes quantity, method of use (e.g. dried cannabis smoked, concentrate vaped, edibles, etc.), frequency, strain, and potency (e.g., THC %, THC/CBD).
Change in problematic cannabis use | Baseline, 2 months, 5 months
  Cannabis Use Disorder Identification Test - Revised (CUDIT-R) will be used to measure problematic cannabis use scores on a scale of 0-32 with higher scores indicating more problematic use.
Change in alcohol consumption | Baseline, 2 months, 5 months
  Alcohol Timeline Followback (TLFB) is a retrospective 30 day calendar method used to collected the number of drinks consumed on each day of the past month. Changes in alcohol consumption will be measured (mL per day).
Change in problematic alcohol use | Baseline, 2 months, 5 months
  Alcohol Use Disorder Identification Test (AUDIT) will be used to measure problematic alcohol use on a scale of 0-40 with higher scores indicating more problematic use.

SECONDARY OUTCOMES:
Readiness to change substance use | Baseline
  A contemplation ladder will be used to assess willingness to change alcohol and/or cannabis use to explore if readiness to change influences engagement with treatment and outcomes.
Change in overall substance use | Baseline, 2 months, 5 months
  The WHO Alcohol, Smoking, and Substance Involvement Screening Test (WHO-ASSIST) will measure substance use risk scores to account for problematic use other than cannabis use. Scores range from 0-39 for each substance with higher scores indicating more severe risk associated with use.
Change in psychotic symptom severity | Baseline, 2 months, 5 months
  The Positive and Negative Symptom Scale (PANSS) will measure psychotic symptom severity across positive, negative and general domains. Positive and negative symptomatology score both range from 7 to 49, and a general psychopathology score range from 16 to 112, with a total score range from 30 to 210. Higher scores indicate higher severity of symptoms.
Change in severity of illness | Baseline to 5 months
  Clinical Global Impression Scale - Severity (CGI-S) at baseline and then the complementary scale for follow-up the Clinical Global Impression Scale - Improvement (CGI-I) will measure changes from baseline in participants overall illness severity at 5 months, The CGI-S, a 7-point clinician rated Likert scale that measures individuals' overall illness severity relative those who the clinician has experienced with the same diagnosis (ranging from 1 = Normal, not at all ill to 7 = Extremely ill). The CGI-I is based on the CGI-S rating and is a 7-point clinician rated Likert scale ranging from 1 = Very much improved to 7 = Very much worse.
Change in functioning | Baseline, 2 months, 5 months
  The World Health Organization Disability Assessment Schedule 2 (WHODAS 2.0) will measure functioning across cognitive, mobility, self-care, getting along, life activities, and participation domains. Total scores range from 40 to 180 with higher scores indicating worse functioning.
Change in depression symptoms | Baseline, 2 months, 5 months
  Calgary Depression Scale for Schizophrenia (CDSS) will measure the level of depression based on symptoms seen in people with a schizophrenia spectrum disorder. Total scores range from 0-27 with higher scores indicating more severe depression.
Change in anxiety symptoms | Baseline, 2 months, 5 months
  Beck Anxiety Inventory (BAI) will measure anxiety symptoms on a scale of 0-63 with higher scores indicating more severe anxiety.
Change in verbal learning | Baseline, 2 months, 5 months
  The California Verbal Learning Test - Third Edition (CVLT3) will be used to measure changes in verbal learning index scores from baseline to 6 months. The CVLT3 measures episodic verbal learning including verbal learning, immediate memory, and delayed memory. The CVLT3 yields three index scores of overall verbal learning and memory performance using a mean of 100 and a standard deviation (SD) of 15 points. The scores range from 40-160, which is 4 SDs below and above the mean.
Change in processing speed | Baseline, 2 months, 5 months
  Trial Making Test A (TMT-A) will measure processing speed in recorded time taken to complete the task for drawing a line between numbers in order. Recorded test time more than 78 seconds indicates deficits in processing speed.
Change in executive functioning | Baseline, 2 months, 5 months
  Trail Making Test B (TMT-B) will be used to measure changes in recorded time taken to complete the task. The assessment requires participant to draw a continuous line between circles containing letters and numbers in the correct ascending sequence (i.e., 1-A-2-B-3-C, etc.). Recorded test time more than 180 seconds indicates deficits in executive functioning.
Change in attention | Baseline, 2 months, 3 months
  The digit vigilance test will measure attention during a rapid visual tracking task. Scores are calculated for the total time and total errors.
Change in social cognition | Baseline, 2 months, 3 months
  The Mayer-Salovey-Caruso Emotional Intelligence Test (MSCEIT) will provide a social cognition composite score based on four branches of emotional intelligence: perceiving emotions, facilitating thought, understanding emotions, and managing emotions. The average MSCEIT score is 100 with a standard deviation of 115.

CONTACTS AND LOCATIONS:
Overall Officials: Philip G Tibbo, MD, Principal Investigator — Nova Scotia Health Authority
Locations (2):
- Canada (2):
  - Psychosis Intervention Early Recovery program, St. John's, Newfoundland and Labrador
  - Nova Scotia Early Psychosis Program, Halifax, Nova Scotia

IPD SHARING:
Plan to Share IPD: No
IPD will only be shared between the Nova Scotia and Newfoundland sites. Data sharing was not a requirement of the study's funding, and given the small sample size, there is a heightened risk of re-identification of participants. To protect participant confidentiality and adhere to institutional ethics guidelines, data will remain securely stored and will not be made available to external parties.